CLINICAL TRIAL: NCT05086289
Title: Randomized Placebo-controlled Phase 2 Clinical Trial to Evaluate LY3526318 for the Treatment of Chronic Low Back Pain
Brief Title: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17515; H0P-MC-BP02 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3526318 (Experimental): Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period and were switched to placebo once daily for the next 4 weeks of the treatment period.
  Interventions: Drug: LY3526318
- Placebo (Placebo Comparator): Participants received placebo orally, once daily, for 8-weeks treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally
  Arms: LY3526318
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether LY3526318 is efficacious and safe in relieving chronic low back pain (CLBP). This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions for the duration of the study.
* Are at 18 years old or older at the time consent is signed.
* Have a history of low back pain for at least 3 months located between the 12th thoracic vertebra and the lower gluteal folds, with or without radiation.
* Have a history of low back pain as classified by the Quebec Task Force Category 1 through 3.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have fibromyalgia
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Have used a therapeutic injection (botulinum toxin or corticosteroids) in the 3 months prior to starting the washout period.
* Have history of or current compression fracture.
* Have had a recent major trauma (within 6 months of baseline).
* Have a history of low back pain as classified by the Quebec Task Force categories 4 through 11.
* Are using a spinal cord stimulator or dorsal root ganglion stimulator.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or (1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (29):
  - Synexus- Chandler, Chandler, Arizona
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Alliance for Multispecialty Research, LLC Tempe, Tempe, Arizona
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Synexus - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Synexus - US, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Chronic Low Back Pain — https://trials.lillytrialguide.com/en-US/trial/7MucQVESfEAcnl27S8VdfF

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 Milligram (mg) LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period and were switched to placebo once daily for the next 4 weeks of the treatment period.
Period: Overall Study
Arm/Group | 250 Milligram (mg) LY3526318 | Placebo
Started | 105 | 54
Received at Least One Dose of Study Drug (Safety Population Week 1-4) | 105 | 54
Safety Population Week 5-8 (All participants who took at least 1 dose of study drug and who did not discontinue at or prior to week 4.) | 92 | 50
Completed | 90 | 49
Not Completed | 15 | 5
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Non-compliance with study drug | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled or randomized participants who received at least one dose of study drug.
Groups:
- 250 mg LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period and were switched to placebo once daily for the next 4 weeks of the treatment period.
- Total: Total of all reporting groups
Arm/Group | 250 mg LY3526318 | Placebo | Total
Number analyzed (Participants) | 105 | 54 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.00 (13.20) | 54.30 (13.74) | 54.10 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 35 | 101
  Male | 39 | 19 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 15 | 40
  Not Hispanic or Latino | 80 | 39 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 84 | 42 | 126
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 2 | 2 | 4
  United States | 103 | 52 | 155
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  score on a scale | 5.56 (1.57) | 5.79 (1.54) | 5.64 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) at Week 4
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95 percent (%) credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 92 | 50
score on a scale | -1.28 [-1.59 to -0.97] | -0.90 [-1.32 to -0.48]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.38, 95% CI 2-sided [-0.89 to 0.13] — Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline for Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 87 | 47
score on a scale | -1.47 [-1.82 to -1.12] | -1.20 [-1.67 to -0.73]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.28, 95% CI 2-sided [-0.85 to 0.30] — Posterior mean difference with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline on the Roland Morris Disability Questionnaire (RMDQ)
Description: The RMDQ is a simple, sensitive, and reliable method to measure disability in patients with back pain that consists of 24 statements relating to the person's perceptions of back pain and associated disability based on physical ability/activity, sleep/rest, psychosocial, household management, eating, and pain frequency. Participants are asked if they feel the statement is descriptive of their own circumstance on that day. The total score is obtained by counting the number of ''Yes'' responses, ranging from: 0 = no disability to 24 = maximal disability.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: All enrolled who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 52
score on a scale | -2.03 [-2.82 to -1.25] | -1.42 [-2.49 to -0.36]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.62, 95% CI 2-sided [-1.91 to 0.68] — Posterior mean difference with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline on the Roland Morris Disability Questionnaire (RMDQ)
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: All enrolled who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 49
score on a scale | -2.55 [-3.37 to -1.71] | -1.37 [-2.49 to -0.25]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -1.17, 95% CI 2-sided [-2.54 to 0.18] — Posterior mean difference with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of Change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7 where, 1=very much better, and 7=very much worse.
  Posterior mean, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 52
score on a scale | 3.13 [2.94 to 3.31] | 3.25 [2.99 to 3.50]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.12, 95% CI 2-sided [-0.44 to 0.19] — Posterior mean difference with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of Change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1 = very much better, and 7 = very much worse.
  Posterior mean, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 49
score on a scale | 3.00 [2.76 to 3.24] | 3.26 [2.93 to 3.59]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.26, 95% CI 2-sided [-0.67 to 0.14] — Posterior mean difference with 95% credible interval is reported

7. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 92 | 50
score on a scale | -1.45 [-1.79 to -1.10] | -0.97 [-1.43 to -0.50]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.48, 95% CI 2-sided [-1.05 to 0.09] — Posterior mean difference with 95% credible interval is reported

8. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 87 | 47
score on a scale | -1.69 [-2.09 to -1.28] | -1.18 [-1.72 to -0.64]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.51, 95% CI 2-sided [-1.17 to 0.16] — Posterior mean difference with 95% credible interval is reported

9. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0=no pain, and 100=worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 52
score on a scale | -14.84 [-18.65 to -10.99] | -9.89 [-14.97 to -4.80]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -4.95, 95% CI 2-sided [-11.07 to 1.27] — Posterior mean difference with 95% credible interval is reported

10. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: as for outcome 9
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 49
score on a scale | -19.50 [-23.74 to -15.30] | -14.72 [-20.39 to -9.00]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -4.78, 95% CI 2-sided [-11.73 to 2.15] — Posterior mean difference with 95% credible interval is reported

11. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Question 1 asks time to fall asleep and it is reported in 5-point timeframe categories. Question 2 asks average hours of sleep. In the remaining 10 questions participants report how often a sleep symptom or problem was present on a scale ranging from '0=all of the time' to '5=none of the time.' MOS Sleep scale dimension scores range from 0 to 100 with lower score indicating improvement, except for the dimension of sleep adequacy, where higher scores indicate improvement. Here, the average hours of sleep (i.e., Question 2) is reported as the average number of hours slept each night during the past week (range 0 to 24 hours). Higher number of hours slept indicates improvement.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 52
Hours per night | 0.11 [-0.09 to 0.32] | 0.24 [-0.04 to 0.52]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.13, 95% CI 2-sided [-0.46 to 0.21] — Posterior mean difference with 95% credible interval is reported

12. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 49
Hours per night | 5.04 [0.08 to 9.95] | 3.52 [-2.96 to 10.02]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 1.52, 95% CI 2-sided [-6.20 to 9.20] — Posterior mean difference with 95% credible interval is reported

13. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score using the United States algorithm. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health: 0=a health state equivalent to death, and 1=perfect health.
  Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 52
score on a scale | 0.02 [-0.02 to 0.06] | 0.01 [-0.04 to 0.07]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.00, 95% CI 2-sided [-0.06 to 0.07] — Posterior mean difference with 95% credible interval is reported

14. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: as for outcome 13
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 49
score on a scale | 0.05 [-0.00 to 0.10] | 0.03 [-0.04 to 0.10]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.02, 95% CI 2-sided [-0.05 to 0.10] — Posterior mean difference with 95% credible interval is reported

15. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: Total amount of rescue medication use as measured by average daily dosage. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg per day (mg/day)
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 92 | 50
mg per day (mg/day) | 229.99 [148.57 to 311.19] | 188.27 [75.50 to 300.88]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 41.72, 95% CI 2-sided [-95.92 to 179.76] — Posterior mean difference with 95% credible interval is reported

16. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: as for outcome 15
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg per day (mg/day)
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 87 | 47
mg per day (mg/day) | 237.79 [144.40 to 332.42] | 228.06 [99.15 to 357.46]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 9.73, 95% CI 2-sided [-151.11 to 170.52] — Posterior mean difference with 95% credible interval is reported

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: All participants under the safety population for week 1-4 and week 5-8. Gender specific events only occurring in male or female participants have had the number of participants at Risk adjusted accordingly.
Groups:
- 250 mg LY3526318 Week 1 to 4: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period (Week 1-4).
- 250 mg LY3526318/Placebo Week 5 to 8: Participants who received 250 mg of LY3526318 in the first 4 weeks were switched to receive placebo once daily for the next 4 weeks of the treatment period (Week 5-8).
- Placebo Week 1 to 4: Participants received placebo orally, once daily, for week 1 to 4 of treatment period.
- Placebo Week 5 to 8: Participant from Week 1-4 continued to receive placebo orally, once daily, for week 5 to 8 of treatment period.
Arm/Group | 250 mg LY3526318 Week 1 to 4 | 250 mg LY3526318/Placebo Week 5 to 8 | Placebo Week 1 to 4 | Placebo Week 5 to 8
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/92 | 0/54 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/105 | 0/92 | 0/54 | 0/50
Other Adverse Events (participants affected / at risk) | 36/105 | 14/92 | 19/54 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg LY3526318 Week 1 to 4 (N=105) | 250 mg LY3526318/Placebo Week 5 to 8 (N=92) | Placebo Week 1 to 4 (N=54) | Placebo Week 5 to 8 (N=50)
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 250 mg LY3526318 Week 1 to 4 (N=105) | 250 mg LY3526318/Placebo Week 5 to 8 (N=92) | Placebo Week 1 to 4 (N=54) | Placebo Week 5 to 8 (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/66 | 0 | 2/35 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal distentation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Vaginal discharge*a (Reproductive system and breast disorders) | 1/66 | 0 | 0/35 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatobiliary scan abnormal (Investigations) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT05086289/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT05086289/SAP_003.pdf